CLINICAL TRIAL: NCT02538614
Title: A Phase 1b/2 Study of Idelalisib in Combination With BI 836826 in Subjects With Chronic Lymphocytic Leukemia
Brief Title: Study of Idelalisib in Combination With BI 836826 in Participants With Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-312-1579
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Results first posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — idelalisib; BI 836826

STUDY DESIGN:
Intervention Model Description: Phase 1b: sequential assignment, Phase 2: parallel assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1b: Idelalisib + BI 836826 (Experimental): Participants will receive escalating dose of idelalisib at dose levels, 50 mg, 100 mg, and 150 mg + BI 836826 10 mg on Day 8, 50 mg on Day 9 and Day 15, and 100 mg on Day 22, every 2 weeks through Week 18, and every 4 weeks through Week 46. 2 dose combinations (highRP2D and lowRP2D) will be determined for further evaluations in Phase 2.
  Interventions: Drug: Idelalisib; Drug: BI 836826
- Phase 2 Idelalisib + BI 836826 (Experimental): Participants will be randomly assigned to receive 1 of the 2 dose combinations selected from Phase 1b.
  Interventions: Drug: Idelalisib; Drug: BI 836826

INTERVENTIONS:
Drug: Idelalisib — Tablets administered orally twice daily
  Other Names: GS-1101; CAL-101; Zydelig®
Drug: BI 836826 — Intravenous administration as a rate-controlled infusion

SUMMARY:
This study consists of 2 parts: Phase 1b and Phase 2. Phase 1b will evaluate the safety and tolerability of the combination of idelallisib with the anti-CD37 monoclonal antibody BI 836826 in participants with relapsed/refractory chronic lymphocytic leukemia (R/R CLL), and establish the high recommended Phase 2 combination dose (highRP2D) as well as an alternate lower recommended Phase 2 combination dose (lowRP2D). Phase 2 will determine the rates of complete response (CR) and of minimal residual disease (MRD) negativity with the combination at the highRP2D and the lowRP2D in participants with R/R CLL.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of B-cell CLL, established according to International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria and having received at least 2 prior treatment regimens
* CLL that warrants treatment
* Clinically quantifiable disease burden defined as:

  * For Phase 1b individuals: absolute lymphocyte count (ALC) > 5000/μL in peripheral blood.
  * For Phase 2 individuals either:

    * At least 1 node ≥ 2 cm on computed tomography (CT) or magnetic resonance imaging (MRI) or
    * bone marrow exam is performed at screening and demonstrates quantifiable CLL.
* Discontinuation of all cytotoxic chemotherapy and anti-CD20 antibody therapy for ≥ 4 weeks, alemtuzumab for ≥ 8 weeks, targeted therapy for ≥ 2 weeks, and investigational therapy for ≥ 3 weeks before enrollment (Phase 1b) or randomization (Phase 2). For individuals with relapsed CLL most recently treated with B-cell receptor (BCR) pathway inhibitors who, in the opinion of the investigator, will not tolerate waiting 3 weeks, a washout period of > 5 half-lives is allowed. If on a systemic corticosteroid, the dose must be stable for the previous 4 weeks.
* Eastern Cooperative Oncology Group (ECOG) score of ≤ 2

Key Exclusion Criteria:

* Known histological transformation from CLL to an aggressive lymphoma (ie, Richter transformation)
* Known presence of myelodysplastic syndrome
* History of a non-CLL malignancy except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate-specific antigen for ≥ 1 year prior to enrollment, other adequately treated Stage 1 or 2 cancer currently in complete remission, or any other cancer that has been in complete remission for ≥ 2 years.
* Evidence of ongoing systemic bacterial, fungal, or viral infection at the time of enrollment
* Ongoing drug-induced liver injury, chronic active hepatitis C (HCV), chronic active hepatitis B (HBV), alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, or portal hypertension.
* History of drug-induced pneumonitis
* Ongoing inflammatory bowel disease
* Ongoing alcohol or drug addiction
* History of prior allogeneic bone marrow progenitor cell or solid organ transplantation
* Ongoing systemic immunosuppressive therapy other than corticosteroids
* History of prior therapy with any phosphatidylinositol 3-kinase (PI3K) inhibitor (including idelalisib), or any anti-CD37 agent
* Ongoing infection with, or treatment or prophylaxis for, CMV within the past 28 days.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-12-29 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (2):
- United States (2):
  - Ohio State University, Columbus, Ohio
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 29 December 2015. The last study visit occurred on 05 July 2017.
Pre-assignment Details: 5 participants were screened. Due to the early study termination, phase 2 was not initiated. Enrollment to this study was closed during Phase 1b. The 2 enrolled participants were allowed to remain on the study.
Groups:
- Phase 1b: Idelalisib + BI 836826: Idelalisib 50 mg tablet was administered orally twice daily each day until the end of treatment. BI 836826 was administered intravenously as a rate-controlled infusion. An initial dose of 10 mg was administered on Day 8. Doses of 50 mg were administered on Day 9 and Day 15. The full assigned dose of 100 mg was administered on Day 22, every 2 weeks thereafter through Week 18, and every 4 weeks thereafter through Week 46.
Period: Overall Study
Arm/Group | Phase 1b: Idelalisib + BI 836826
Started | 2
Completed | 0
Not Completed | 2
Not completed — Progressive Disease | 2

BASELINE CHARACTERISTICS:
Population: The All Enrolled Analysis Set included all participants who were enrolled in the study.
Arm/Group | Phase 1b: Idelalisib + BI 836826
Number analyzed (Participants) | 2
Age, Customized [Count of Participants; unit: Participants]
  >= 65 Years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race-Data not reported | NA — Data are not reported for participant confidentiality reasons.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity-Data not Reported | NA — Data are not reported for participant confidentiality reasons.
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Percentage of Participants Experienced Dose Limiting Toxicities (DLTs) During the First 7 Weeks of Study Therapy
Description: DLTs refer to toxicities experienced during the final 6 weeks of 7-week study treatment that have been judged to be clinically significant and related to study treatment. Events occurring during the initial 7-day idelalisib monotherapy run-in period and resolving by Day 8 were not included.
Time Frame: Up to 7 weeks
Population: Due to early study termination this outcome measure was not assessed.
Arm/Group | Phase 1b: Idelalisib + BI 836826
Number analyzed (Participants) | 0

2. Primary Outcome: For Phase 2: Complete Response Rate (CRR)
Description: CRR was defined as the percentage of participants who achieve a complete response (CR). CR was defined as the complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease.
Time Frame: Up to 18 months
Population: Due to early study termination this outcome measure was not assessed.
Groups:
- Phase 2: Idelalisib + BI 836826: Phase 1b-Idelalisib 50 mg tablet was administered orally twice daily each day until the end of treatment. BI 836826 was administered intravenously as a rate-controlled infusion. An initial dose of 10 mg was administered on Day 8. Doses of 50 mg were administered on Day 9 and Day 15. The full assigned dose of 100 mg was administered on Day 22, every 2 weeks thereafter through Week 18, and every 4 weeks thereafter through Week 46.
  Phase 2 did not occur.
Arm/Group | Phase 2: Idelalisib + BI 836826
Number analyzed (Participants) | 0

3. Primary Outcome: For Phase 2: Minimal Residual Disease (MRD) Negativity Rate in Bone Marrow by Week 50
Description: MRD defined as the percentage of participants with MRD < 10^-4, assessed by flow cytometry in bone marrow, achieved by Week 50.
Time Frame: Week 50
Population: Due to early study termination this outcome measure was not assessed.
Arm/Group | Phase 2: Idelalisib + BI 836826
Number analyzed (Participants) | 0

4. Secondary Outcome: Phase 1b: Percentage of Participants Experienced DLTs During the Treatment Period
Description: as for outcome 1
Time Frame: Up to 18 months
Population: Due to early study termination this outcome measure was not assessed.
Arm/Group | Phase 1b: Idelalisib + BI 836826
Number analyzed (Participants) | 0

5. Secondary Outcome: For Phase 1b and Phase 2: Number of Participants Experiencing Any Serious Adverse Events (SAE)
Description: An SAE is defined as an event that, at any dose, results in the following: death, life-threatening, in-patient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, a congenital anomaly/birth defect or a medically important event or reaction.
Time Frame: Up to 18 months
Population: The Safety Analysis Set included all participants who received at least 1 dose of any study drug, with treatment group designated according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b and 2: Idelalisib + BI 836826: Phase 1b-Idelalisib 50 mg tablet was administered orally twice daily each day until the end of treatment. BI 836826 was administered intravenously as a rate-controlled infusion. An initial dose of 10 mg was administered on Day 8. Doses of 50 mg were administered on Day 9 and Day 15. The full assigned dose of 100 mg was administered on Day 22, every 2 weeks thereafter through Week 18, and every 4 weeks thereafter through Week 46.
  Phase 2 did not occur.
Arm/Group | Phase 1b and 2: Idelalisib + BI 836826
Number analyzed (Participants) | 2
Participants | 2

6. Secondary Outcome: For Phase 1b and Phase 2: Number of Participants Who Permanently Discontinued Study Treatment Due to an Adverse Event
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal product, which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. The severity of AEs was graded using the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.
Time Frame: Up to 18 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b and 2: Idelalisib + BI 836826
Number analyzed (Participants) | 2
Participants | 0

7. Secondary Outcome: For Phase 2: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants achieving a complete response (CR) or partial response (PR). CR was defined as the complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease. PR was defined as a ≥ 50% reduction in the sum of the products of the longest perpendicular diameters of all index lesions, with no new lesions.
Time Frame: Up to 18 months
Population: Due to early study termination this outcome measure was not assessed.
Arm/Group | Phase 2: Idelalisib + BI 836826
Number analyzed (Participants) | 0

8. Secondary Outcome: For Phase 2: Duration of Complete Response (DCR)
Description: DCR was defined as the interval from the first documentation of CR to the earlier of the first documentation of definitive disease progression or death from any cause. CR was defined as the complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease.
Time Frame: Up to 18 months
Population: Due to early study termination this outcome measure was not assessed.
Arm/Group | Phase 2: Idelalisib + BI 836826
Number analyzed (Participants) | 0

9. Secondary Outcome: For Phase 2: Duration of Response (DOR)
Description: DOR was defined as the interval from the first documentation of CR or PR to the earlier of the first documentation of definitive disease progression or death from any cause. CR was defined as the complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease. PR was defined as a ≥ 50% reduction in the sum of the products of the longest perpendicular diameters of all index lesions, with no new lesions.
Time Frame: Up to 18 months
Population: Due to early study termination this outcome measure was not assessed.
Arm/Group | Phase 2: Idelalisib + BI 836826
Number analyzed (Participants) | 0

10. Secondary Outcome: For Phase 2: Progression-Free Survival (PFS)
Description: PFS was defined as the interval from randomization to the earlier of the first documentation of definitive disease progression or death from any cause. Definitive disease progression was defined as evidence of any new disease, worsening of index lesions, spleen or liver, or non-index disease, decrease in platelet count or hemoglobin that is attributable to chronic lymphocytic leukemia (CLL) or more than 4 weeks after the discontinuation of idelalisib: an increase in the number of blood lymphocytes by 50% or more.
Time Frame: Up to 18 months
Population: Due to early study termination this outcome measure was not assessed.
Arm/Group | Phase 2: Idelalisib + BI 836826
Number analyzed (Participants) | 0

11. Secondary Outcome: For Phase 2: Overall Survival (OS)
Description: OS was defined as the interval from the randomization to the date of death from any cause.
Time Frame: Up to 18 months
Population: Due to early study termination this outcome measure was not assessed.
Arm/Group | Phase 2: Idelalisib + BI 836826
Number analyzed (Participants) | 0

12. Secondary Outcome: For Phase 2: MRD Negativity Rate in Blood at Any Time
Description: MRD negativity rate in blood was defined as the percentage of participants with MRD < 10^-4, assessed by flow cytometry in blood, at any time on study.
Time Frame: Up to 18 months
Population: Due to early study termination this outcome measure was not assessed.
Arm/Group | Phase 2: Idelalisib + BI 836826
Number analyzed (Participants) | 0

13. Secondary Outcome: For Phase 2: MRD Negativity Rate in Bone Marrow at Any Time
Description: MRD negativity rate in bone marrow was defined as the percentage of participants with MRD < 10^-4, assessed by flow cytometry in bone marrow, at any time on study.
Time Frame: Up to 18 months
Population: Due to early study termination this outcome measure was not assessed.
Arm/Group | Phase 2: Idelalisib + BI 836826
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first dose date to study termination (up to approximately 18 months)
Description: The Safety Analysis Set included all participants who received at least 1 dose of any study drug, with treatment group designated according to the actual treatment received.
Arm/Group | Phase 1b: Idelalisib + BI 836826
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Idelalisib + BI 836826 (N=2)
Upper respiratory tract infection (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Idelalisib + BI 836826 (N=2)
Anaemia (Blood and lymphatic system disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Infusion site bruising (General disorders) | 1
Localised oedema (General disorders) | 1
Oedema (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Rhinovirus infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT02538614/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT02538614/SAP_001.pdf